CLINICAL TRIAL: NCT06691243
Title: Evaluation Of Semaglutide Safety and Tolerability in Adults With Cocaine Use Disorder With and Without HIV
Brief Title: Evaluation Of Semaglutide in Adults With Cocaine Use Disorder With and Without HIV
Acronym: STAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sarah Kattakuzhy, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00112237; 75N90024C00036 (Other: NIH Clinical Center)
Record Dates: First submitted 2024-11-06; First posted 2024-11-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cocaine Use Disorder; HIV
Keywords: semaglutide; GLP-1; cocaine use disorder
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Once weekly injection of semaglutide
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Once weekly injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — The initial dose will be semaglutide 0.25mg which, if tolerated, will be escalated to 0.5mg. Escalation will continue to 1.0 mg and afterwards to 2.0 mg. The highest possible dose will be 2.0mg semaglutide.
  Other Names: Wegovy; Ozempic
  Arms: Semaglutide
Drug: Placebo — Patients randomized to placebo arm will receive placebo injection every week.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to find out if semaglutide is safe and well tolerated in adults with cocaine use disorder who do and do not have human immunodeficiency virus (HIV). Participants will complete a screening process and if you are able to participate, you will be assigned to one of two treatment groups: semaglutide or placebo.

Participants will:

* Visit the clinic once a week for semaglutide or placebo injections
* Visit the clinic once every two weeks for labwork, assessments and/or surveys
* If consented to optional MRI's, complete two MRI's

DETAILED DESCRIPTION:
STAC is a 16-week, double-blind, placebo-controlled, pilot, dose-escalation study that aims to determine the dose of semaglutide that is safe and tolerable in individuals with cocaine use disorder, including those with and without HIV; whether semaglutide improves drug use outcomes for cocaine use; and whether semaglutide improves cardiac and inflammatory biomarkers. Interested participants will be consented and screened, and after screening process is completed, all eligible participants who desire to continue with the study will be randomized either to semaglutide injections or placebo injections. Participants will receive semaglutide or placebo injections once a week from Day 0 through Week 16, and a final assessment will be completed at Week 16. Study visits will also intermittently complete labwork, medical examinations, clinical assessments and surveys.

Participants who consent to the optional MRI visits, will also complete MRI's at two timepoints: once before starting the study medication and once near Week 16.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Meet criteria for CUD according to the Diagnostic and Statistical Manual Version 5
3. Used cocaine at least 7 out of the past 14 days
4. Body Mass Index between 20 - 50 kg/m2
5. English proficiency
6. In people of childbearing potential, agree to use an acceptable method of birth control

Exclusion Criteria:

1. Triglycerides > 500 mg/dL
2. History of gall bladder disease
3. Personal or family history of medullary thyroid carcinoma, or patients with a history of Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
4. History of diabetic retinopathy
5. Being prescribed glucose-lowering medications
6. An estimated glomerular filtration rate of less than 45 ml/min
7. Lifetime history of taking semaglutide or other GLP-1 RAs
8. Current suicidal ideation or suicide attempts within the past 24 months
9. Present diagnosis of diabetes mellitus OR screening hemoglobin A1C >/= 6.5
10. Use of weight-lowering medications
11. History of gastric bypass surgery
12. History of myocardial infarction or stroke within the past 12 months
13. Pregnant, breastfeeding, or the patient intends to become pregnant during the next four months
14. Any contraindicated medical issues identified by the study investigators
15. Risk of conditions that are under Warning and Precautions section of OZEMPIC and WEGOVY including but not limited to known history or current report of clinically relevant hypoglycemia, gastroparesis, or pancreatic disease.
16. Calcitonin value equal to or above 50 ng/L
17. If completing the MRI portion of the study: claustrophobia or physical issues preventing MRI scan
18. If completing the MRI portion of the study: presence of a metal device in the body (e.g. pacemaker. Infusion pump, aneurysm clip, metal prosthesis or plate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of semaglutide in patients with cocaine use disorder (CUD) with and without HIV | 16 weeks
  Number of Grade 3 and 4 adverse effects reported by patients at any time after Day 0
Tolerability of semaglutide in patients with cocaine use disorder (CUD) with and without HIV | 16 weeks
  Dose of semaglutide the patient tolerates regardless of the presence of adverse effects

SECONDARY OUTCOMES:
Determine if semaglutide improves cocaine use frequency in people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in cocaine use frequency via timeline followback method. The higher the frequency of cocaine use, the worse the outcome.
Determine if semaglutide reduces cocaine use in people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose of mean dollar-amount patients spent on cocaine during the past 7 days. The higher the amount, the worse the outcome.
Determine if semaglutide reduces cocaine use in people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in presence of cocaine metabolite detected on urine drug-screen results.
Determine if semaglutide reduces cocaine craving for people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Cocaine Craving Questionnaire Brief (CCQ-Brief). Minimum score= 8 (minimal craving). Maximum score= 56 (extreme craving). The higher the score, the worse the outcome.
Determine if semaglutide reduces drug use severity for people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on the Drug Abuse Screening Test (DAST). Minimum Value= 0 (No problems with drug abuse or dependence. Maximum Value= 10 ( severe drug-related problems). The higher the score, the worse the outcome.
Determine if semaglutide reduces risk taking behavior in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Balloon Analogue Risk Task (BART). Minimum score= 0 (no risk taking). Maximum: Variable, it can go up to 500-1000. Higher Scores= Higher risk taking behavior.
Determine if semaglutide reduces impulsiveness in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Barratt Impulsiveness Scale (BAS-11) Minimum score: 30, Maximum score: 120. Higher score equals high impulsivity.
Determine if semaglutide reduces compulsivity in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Obsessive-Compulsive Cocaine Use Scale. Minimum score: 0 (no symptoms), Maximum Score: 32. Higher score = greater severity of obsessive-compulsive symptoms related to cocaine use. The higher the score, the worse the outcome.
Determine if semaglutide impacts depression in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Patient Health Questionnaire-9 (PHQ-9). Minimum score: 0 (no depressive symptoms). Maximum score: 27 (severe depression). Higher score indicates worse outcome.
Determine if semaglutide impacts anxiety in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Generalized Anxiety Disorder-7 (GAD-7). Minimum score= 0 (no anxiety symptoms). Maximum= 21 (severe anxiety) Higher score indicates worse outcome.
Determine if semaglutide impacts anhedonia in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Snaith-Hamilton Pleasure Scale (SHAPS). Minimum score=0 (no anhedonia). Maximum score=14 (severe anhedonia). The higher the score, the worse the outcome
Determine if semaglutide impacts sleep in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on Pittsburgh Sleep Quality Index (PSQI). Minimum score= 0 (good sleep quality). Maximum= 21 (poor sleep quality). The higher the score, the worse the outcome.
Determine if semaglutide impacts sexual desire in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on the Sexual Desire Inventory (SDI).- Minimum score= 0 (no sexual desire). Maximum score= 60 (high sexual desire). The lower the score, the worse the outcome.
Determine if semaglutide impacts food cravings in people with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in score on the General Trait Food Cravings Questionnaire (G-FCQ-T). Minimum score = 0 (no food cravings). Maximum score =7 (high frequency and intensity of cravings). The lower the score, the worse the outcome.
Determine if semaglutide changes levels of inflammatory biomarkers in patients with HIV relative to those without HIV | 16 weeks
  Levels of HIV-induced inflammation markers (inflammatory cytokines, IFN-g, TNF, IL-6, IL-8, chemokine, IL18, CD163, Neopterin, beta 2 microglobulin, LPS, sCD14, sCD25, IL12, IL10) before and after s.c. semaglutide
Determine if semaglutide changes levels of clinically relevant cardiovascular biomarkers in patients with HIV relative to those without HIV | 16 weeks
  Levels of cardiovascular biomarkers (levels of high-sensitivity C-reactive protein (CRP), high-sensitivity troponin (hs- hs-TRP), endothelin-1 (ET-1), D-dimer before and after s.c. semaglutide
Determine if semaglutide effects changes in body fat in individuals with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in percent body fat using the InBody scan. The lower the percent body fat, the worse the outcome.
Determine if semaglutide effects body fat distribution in people with CUD with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in body fat distribution. The more central the body fat distribution, the worse outcomes.
Determine if semaglutide effects changes muscle mass in patients with cocaine use disorder, with and without HIV | 16 weeks
  Change from baseline to highest tolerated semaglutide or placebo dose in percent muscle mass using the InBody Scan. The lower the percentage of muscle mass, the worse the outcome.
Determine if s.c. semaglutide produces changes in brain function in patients with cocaine use disorder, with and without HIV | 16 weeks
  Magnetic Resonance Spectroscopy (MRS)will be used to assess whether s.c. semaglutide produces changes in brain metabolite levels; Resting state functional connectivity (RSFC) will be used to assess whether s.c. semaglutide produces changes in brain network function; An Arterial Spin Labeling (ASL) sequence that measures Blood Brain Barrier (BBB) permeability will be used to assess whether s.c. semaglutide produces changes in BBB integrity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute of Human Virology at the University of Maryland School of Medicine, Washington D.C., District of Columbia
  - Institute of Human Virology at the University of Maryland School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD necessary to verify study results
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after study completion.
Access Criteria: Investigators can email the Principal Investigator (PI) with access requests and the PI will judge if the use of data is justified. If the PI deems the research question appropriate, the PI will grant access.